CLINICAL TRIAL: NCT03521557
Title: Gaze and Postural Stability in People With MS: Characterizing Deficits and Response to Treatment
Brief Title: Gaze and Postural Stability in Multiple Sclerosis
Acronym: GPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Multiple Sclerosis Society (Other); Arizona State University (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Lee Dibble, Professor, University of Utah
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IRB_00104298
Record Dates: First submitted 2017-10-27; First posted 2018-05-11 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Multiple Sclerosis; Vertigo; Dizziness; Falls Injury
MeSH Terms: conditions — Multiple Sclerosis; Vertigo; Dizziness

STUDY DESIGN:
Intervention Model Description: 2 group x 3 time interval
Who Masked: Outcomes Assessor
Masking Description: Participants will be assessed at baseline prior to randomization. Once baseline assessments are completed, participants will be randomized to one of 2 study groups. Interventions will occur at a different site than assessments to avoid unmasking. At the post test and follow-up assessment time points, participants will be instructed not to divulge their group assignment to their assessor (the same individual that assessed them at baseline).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gaze and Postural Stability (Experimental): The duration and content of the Gaze and Postural Stability (GPS) intervention is specifically designed to focus on gradually increasing difficulty of gaze and postural stability exercises.
  The target duration of each in clinic visit will be 90 min (15 min of gaze stability exercises, 15 min of postural stability exercises and approximately 60 min for the standard care control intervention with rest interspersed throughout the exercise session.
  Gaze stability exercise will consist of progressive Vestibular-occular training.
  Postural stability exercises will consist of progressive static and dynamic postural training.
  Interventions: Behavioral: Gaze and Postural Stability; Behavioral: Standard Care Control
- Standard Care Control (Active Comparator): The Standard Care Control intervention is specifically designed to be focused on improving overall endurance and lower extremity muscular strength. The target duration of each in clinic visit will be 90 min (30 min of aerobic exercise, 30 min of lower extremity resistance exercises, and 30 min of rest interspersed throughout the exercise session.
  Interventions: Behavioral: Standard Care Control

INTERVENTIONS:
Behavioral: Gaze and Postural Stability — The duration and content of the GPS intervention is specifically designed to focus on gradually increasing difficulty of gaze and postural stability exercises.
  Other Names: GPS
  Arms: Gaze and Postural Stability
Behavioral: Standard Care Control — The Standard Care Control intervention is specifically designed to be focused on improving overall endurance and lower extremity muscular strength.
  Other Names: Standard Care Control (SCC)

SUMMARY:
In order to provide information that will improve therapy, the goals of this project are to determine if persons with MS with complaints of dizziness and at risk for falls can improve their balance and vision stability as a result of a bout of specific treatment. This project seeks to do this by conducting an experiment where people with MS are randomly assigned to a group that practices activities known to help improve inner ear function or a group that practices activities known to improve endurance and strength but that should not change inner ear function. Such a comparison will allow us to gain understanding of how the inner ear system is affected in MS and how it responds to treatment.

DETAILED DESCRIPTION:
A variety of sources of evidence suggest altered vestibular function in people diagnosed with MS (PwMS). These sources of evidence include [a] subjective complaints of dizziness / vertigo, [b] altered subjective visual vertical, [c] altered vestibular evoked myogenic potentials, [d] altered performance on the vestibular dominant components of the sensory organization test, and [e] pilot reports of gaze stabilization deficits during vestibular ocular reflex (VOR) testing from the investigator's research group. These findings suggest vestibular deficits are present in PwMS. Epidemiological studies document cerebellar and brainstem involvement in 23% of PwMS at disease onset, increasing to 82% after longstanding illness. These vestibular deficits contribute to motion sensitivity, dizziness, imbalance, and falls. Regardless, dizziness and falls have a significant negative impact on quality of life. Multiple studies show that falls are a major disabling symptom in MS affecting approximately 75% of PwMS. The high incidence of falls in MS, is an important health concern due to its associations with injury-related morbidities, mortality and financial costs.

The vestibular pathways responsible for gaze and postural stability, as well as sensory integration reside in the brainstem, cerebellum and spinal cord. Demyelination of the pathways involving the vestibular nuclei complex within the brainstem and cerebellum adversely affect angular vestibulo-ocular reflex,vestibulo-spinal reflex function and sensory integration in PwMS. While evidence reports impairments in posturography and otolith mediated responses (vestibular evoked myogenic potentials), the responses mediated by the semicircular canal end organs and vestibular pathways have not been examined. Specifically, the learning and retention of gaze and postural stability as a result of task specific training program has not been studied in a well controlled clinical trial.

This proposal seeks to examine gaze and postural stability outcomes utilizing outcome measures that span the World Health Organization's International Classification of Function, Disability, and Health. Following completion of the baseline examination, PwMS will be randomized to one of two interventions: An Experimental Gaze and Postural Stability Training Group (GPS) or a Standard Care Aerobic Exercise Control Group (SCA). The two groups differ only by the presence of the GPS program in the experimental group. Both groups will participate in supervised exercise 3 times per week for 6 weeks followed by a post intervention testing period . After one month of no training, both groups will be brought back for a final follow-up examination to determine the retention of any training induced changes.

ELIGIBILITY:
Inclusion Criteria:

* Neurologist-diagnosed, clinically definite MS
* Expanded Disability Severity Scale (EDSS) score of less than 6.0
* Current complaints of dizziness (DHI > 0)
* At risk of falls (determined by > 2 falls in past year or Dynamic Gait Index <19 or Activity Specific Balance Confidence Scale <80
* Ability to tolerate repetitive 5 min bouts of angular head motions.

Exclusion Criteria:

* Central or Peripheral Nervous System disorders (other than MS)
* Otologic, Cervical spine, or lower extremity injury in last 12 months
* Exercise or alcohol use in last 48 hours
* Currently taking vestibular suppressant medications
* Peripheral Vestibular Pathology (BPPV, hypofunction, Meniere's disease
* Internuclear Opthalmoplegia
* MS exacerbation within last 8 weeks
* Orthopedic, neurologic, or cognitive comorbidities that would limit participation in the study procedures

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory | At intervention completion (6 weeks)
  Dizziness Handicap Inventory (DHI): The DHI is a self assessment inventory designed to evaluate the self-perceived handicap effects imposed by dizziness or unsteadiness and has documented test-retest and internal consistency reliability in PwMS.[72-76]. The DHI consists of 25 questions subgroup into functional, emotional, and physical components. The total score ranges from 0-100, with higher scores indicating greater handicap. Collected at intervention completion, adjusting for baseline (DHI values collected at baseline assessment, prior to intervention).

SECONDARY OUTCOMES:
Dizziness Handicap Inventory Follow-up | 1-month follow-up post intervention (10 weeks)
  Dizziness Handicap Inventory (DHI): The DHI is a self assessment inventory designed to evaluate the self-perceived handicap effects imposed by dizziness or unsteadiness and has documented test-retest and internal consistency reliability in PwMS.[72-76]. The DHI consists of 25 questions subgroup into functional, emotional, and physical components. The total score ranges from 0-100, with higher scores indicating greater handicap. Collected at 1-month follow-up, adjusting for baseline (DHI values collected at baseline assessment, prior to intervention).
Activity Specific Balance Confidence Scale | At intervention completion (6 weeks) and 1-month follow-up post intervention (10 weeks)
  The Activity Specific Balance Confidence Scale (ABC) is a 16-item self-reported measure of balance confidence in performing various activities of daily living. Each question requires an individual to grade his or her self on a scale of 0 to 100 percent for their level of confidence and higher scores indicate greater balance confidence in performing these activities. Collected at intervention completion and 1 month follow-up adjusted for baseline (values collected prior to intervention).
Functional Gait Assessment | At intervention completion (6 weeks) and 1-month follow-up post intervention (10 weeks)
  The Functional Gait Assessment (FGA) is a 10-item measure that examines dynamic stability during various walking tasks on a marked 6-m (20-ft) length and 12-inch wide walkway. Each item is rated from 0-3 with higher scores indicating better dynamic stability. Tasks within the FGA require head and / or body motion during walking activities which will be assessed using body-worn 3D accelerometers. Collected at intervention completion and 1-month follow-up adjusting for baseline (values collected at baseline assessment).
Mini-BEST test | At intervention completion (6 weeks) and 1-month follow-up post intervention (10 weeks)
  the 14-item Mini-BESTest which includes four sections (anticipatory postural adjustments, reactive postural responses, sensory orientation, and stability in gait) relevant to postural control and stability in MS.[37] The maximum possible score is 28 with higher scores indicating better balance. Tasks within the Mini-BEST test require head and/ or body motion, which will be assessed using body-worn 3D accelerometers. Collected at intervention completion and 1-month follow-up adjusting for baseline (values collected at baseline assessment).
Dynamic Visual Acuity | At intervention completion (6 weeks) and 1-month follow-up post intervention (10 weeks)
  The Dynamic Visual Acuity (DVA) test is a valid and reliable functional measure of gaze stability that utilizes head rotations representing natural head velocities during daily activities. The variable logMAR is the standard measurement for DVA and is equal to log10x, where x is the minimum angle resolved, in arcmin, with 1 arcmin equal to 1/60°). The better one's visual acuity, the lower one's logMAR score. Collected at intervention completion and 1-month follow-up adjusting for baseline (values collected at baseline assessment).
Passive Angular Vestibulo-ocular Reflex Gain | At intervention completion (6 weeks) and 1-month follow-up post intervention (10 weeks)
  The angular vestibular ocular reflex (aVOR) gain will be calculated as the ratio of the de-saccaded eye velocity Area Under the Curve (AUC) over the head velocity AUC between the onset of the head impulse to the moment when head velocity returns to zero. Collected at intervention completion and 1-month follow-up adjusting for baseline (values collected at baseline assessment).
Compensatory Saccade Frequency | At intervention completion (6 weeks) and 1-month follow-up post intervention (10 weeks)
  The number of Compensatory Saccades (CS) per Head Rotation (CS/HR) will be manually counted per head rotation. Collected at intervention completion and 1-month follow-up adjusting for baseline (values collected at baseline assessment).
Compensatory Saccade Latency | At intervention completion (6 weeks) and 1-month follow-up post intervention (10 weeks)
  The Compensatory Saccade (CS) latency is the duration of time between the onset of head acceleration to onset of first identifiable CS. Collected at intervention completion and 1-month follow-up adjusting for baseline (values collected at baseline assessment).
Gaze Position Error | At intervention completion (6 weeks) and 1-month follow-up post intervention (10 weeks)
  Gaze position error is calculated as the visual target position minus the eye position at the end of the head impulse. Collected at intervention completion and 1-month follow-up adjusting for baseline (values collected at baseline assessment).
Margin of stability | At intervention completion (6 weeks) and 1-month follow-up post intervention (10 weeks)
  the margin of dynamic stability. Margin of dynamic stability characterizes the distance between the base of support and the extrapolated center of mass (a measure which incorporates the position and velocity of the center of mass. Collected at intervention completion and 1-month follow-up adjusting for baseline (values collected at baseline assessment).
Step Latency | At intervention completion (6 weeks) and 1-month follow-up post intervention (10 weeks)
  The step latency will be calculated as the time period between tether release and foot off of the stepping limb. Collected at intervention completion and 1-month follow-up adjusting for baseline (values collected at baseline assessment).
Postural Sway | At intervention completion (6 weeks) and 1-month follow-up post intervention (10 weeks)
  The amount of postural sway during quiet stance on firm, foam, and incline surfaces will be assessed using 3D accelerometers. Collected at intervention completion and 1-month follow-up adjusting for baseline (values collected at baseline assessment).

OTHER OUTCOMES:
Expanded Disability Status Scale | Baseline
  The Expanded Disability Status Scale (EDSS) is a valid and reliable indicator of disability used by referring medical providers in people with multiple sclerosis. Scores range from 0-10, with higher scores indicating greater levels of disability.
Six minute walk test | At intervention completion (6 weeks) and 1-month follow-up post intervention (10 weeks)
  The distance walked in 6 minutes (Six-Minute Walk [6MW]) is a valid and reliable measure of locomotor ability in populations with a variety of chronic diseases including MS. Higher values reflect greater ability. Collected at intervention completion and 1-month follow-up adjusting for baseline (values collected at baseline assessment).
Modified Fatigue Impact Scale | At intervention completion (6 weeks) and 1-month follow-up post intervention (10 weeks)
  Fatigue will be assessed using the abbreviated 5-item version of the Modified fatigue impact scale (MFIS). The scale contains 5 statements that describe how fatigue may impact an individual with MS during the previous 4 weeks. Each item is rated on a 5-point ordinal scale; total scores range from 0 to 20, and lower scores indicating less fatigue. Collected at intervention completion and 1-month follow-up adjusting for baseline (values collected at baseline assessment).
25 foot walk test | At intervention completion (6 weeks) and 1-month follow-up post intervention (10 weeks)
  Patient walking speed will be assessed using a 25 foot walkway. Participants are instructed to walk at their normal pace the length of the walkway while being timed. Collected at intervention completion and 1-month follow-up adjusting for baseline (values collected at baseline assessment).

CONTACTS AND LOCATIONS:
Overall Officials: Lee Dibble, PhD, PT, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Loyd BJ, Saviers-Steiger J, Fangman A, Ballard P, Taylor C, Schubert M, Dibble L. Turning Toward Monitoring of Gaze Stability Exercises: The Utility of Wearable Sensors. J Neurol Phys Ther. 2020 Oct;44(4):261-267. doi: 10.1097/NPT.0000000000000329. PMID 32815892
- [Derived] Loyd BJ, Fangman A, Peterson DS, Gappmaier E, Schubert MC, Thackery A, Dibble L. Rehabilitation to improve gaze and postural stability in people with multiple sclerosis: study protocol for a prospective randomized clinical trial. BMC Neurol. 2019 Jun 10;19(1):119. doi: 10.1186/s12883-019-1353-z. PMID 31179920